CLINICAL TRIAL: NCT07369557
Title: MB-TBS: Mindfulness-Based Theta-Burst Stimulation-A Pilot Study Integrating Mindfulness Training Into Accelerated Neuromodulation Therapy for Depression
Brief Title: Mindfulness Training During Accelerated iTBS for Depression (MB-TBS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Wisconsin, Madison (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Clayton Olash, Medical/Dental Resident, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00148491; R25DA020537 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depression
Keywords: Major Depressive Disorder; Transcranial Magnetic Stimulation; Theta-Burst Stimulation; Mindfulness; Positive Affect; Hedonic Tone
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Training during aiTBS (Experimental)
  Interventions: Behavioral: Guided Mindfulness Practice (Healthy Minds app)

INTERVENTIONS:
Behavioral: Guided Mindfulness Practice (Healthy Minds app) — One guided "Foundation" per day (5-30 minutes) during aiTBS inter-session intervals for five consecutive treatment days; optional additional practices allowed. App analytics (with permission) and self-reports quantify engagement.

SUMMARY:
This NIH-funded single-arm pilot tests the feasibility, acceptability, and preliminary effects of embedding brief guided mindfulness practice (via the Healthy Minds smartphone app) into the inter-session intervals of clinically administered accelerated intermittent theta-burst stimulation (aiTBS) for major depressive disorder (MDD). Participants receive aiTBS as standard clinical care at MUSC; the research intervention is daily guided mindfulness practice during the aiTBS course. Outcomes include feasibility/acceptability, changes in state mindfulness and hedonic tone (Day 0 to Day 5), perceived ease of meditation, trait mindfulness at 4 and 12 weeks, and durability of antidepressant response (PHQ-9) at 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDD and eligible for aiTBS at MUSC
* Already enrolled in aiTBS course at MUSC
* English proficiency
* Smartphone or willingness to use study-provided device

Exclusion Criteria:

* TMS contraindications (e.g., seizure history, implants, pregnancy)
* Concurrent neuromodulation (ECT, VNS)
* Psychotic disorder, bipolar disorder, active substance use disorder, high suicide risk
* Unable/unwilling to engage in mindfulness or complete questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Guided Mindfulness Practice During aiTBS (Adherence Rate) | Day 0 to Day 5
  Proportion of participants who complete ≥1 Healthy Minds Foundation guided practice on each of the five aiTBS treatment days. Calculated as: number completing all five days ÷ total enrolled. Higher values indicate better feasibility.
Tolerability of Guided Mindfulness Practice During aiTBS (Adverse Events) | Day 0 to Day 5
  Number and severity of meditation-related adverse events recorded via participant report and study staff observation. Higher values indicate worse tolerability.

SECONDARY OUTCOMES:
Change in State Mindfulness (Toronto Mindfulness Scale Total Score) | Day 0 to Day 5
  Change in Toronto Mindfulness Scale (TMS) total score from baseline to Day 5. Higher scores indicate greater state mindfulness.
Change in Hedonic Tone (Snaith-Hamilton Pleasure Scale Total Score) | Day 0 to Day 5
  Change in Snaith-Hamilton Pleasure Scale (SHAPS) total score from baseline to Day 5. Lower scores indicate improved hedonic tone.
Change in Perceived Ease of Meditation (0-10 Rating) | Day 0 to Day 5
  Change in meditation ease rating on a 0-10 numeric scale (0 = not at all easy; 10 = extremely easy). Higher scores indicate greater perceived ease.
Change in Trait Mindfulness (CAMS-R Total Score) | Baseline to Week 12 (with Week-4 assessment)
  Change in Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) total score from baseline to Week 12. Higher scores indicate greater trait mindfulness.
Durability of Antidepressant Response (Percent Change in PHQ-9) | Baseline to Week 4
  Percent change in PHQ-9 total score from baseline to Week 4. Lower scores indicate improvement
Meditation Engagement (App Analytics and Self-Report) | Day 0 to Week 12
  Engagement with the Healthy Minds app measured by total minutes practiced, number of Foundations completed, and cumulative meditation minutes. Higher values indicate greater engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Olash, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina (MUSC), Brain Stimulation Laboratory Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Within 12 months of study completion